CLINICAL TRIAL: NCT00302497
Title: 12 Month, Prospective, Randomised, Open-Label Comparative Study to Evaluate the Protection of Kidney Function by Basiliximab in a CNI-Free Regimen in Newly Kidney Transplanted Patients (Three Months Post-Transplant) Who Are Recipient of One Kidney From Expanded Donor Criteria (UNOS Criteria)
Brief Title: EXTEND Protocol for Transplanted Patient to Evaluate Kidney Function
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCHI621ACA07
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2007-04-12 (Estimated); Status verified 2006-02

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Basiliximab

INTERVENTIONS:
Drug: basiliximab

SUMMARY:
The long-term use of calcineurin inhibitors in the maintenance phase after kidney transplantation is associated with typical adverse effects, such as potential contribution to progressive impairment of renal function, hypertension, and metabolic abnormalities.

This 15 month study with a safety follow up is undertaken to evaluate the potential benefit of an alternative treatment strategy to the chronic use of CNI. It will establish, through a comparative design, the superior protection of kidney function provided by chronic usage of basiliximab over tacrolimus early post-transplantation using EDC kidneys.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients aged 40 to 75 years with a viable graft
* patients who are recipients of a primary or secondary graft from a cadaveric expanded donor criteria
* patients who had no change of immunosuppressor two weeks prior to baseline
* patients who had no acute rejection four weeks prior to baseline
* patients who are willing and capable of giving written informed consent for study participation
* females of childbearing potential must have a negative serum pregnancy test within 7 days prior to baseline.Effective contraception must be used during the trial and for 6 weeks following discontinuation of the study medication, even where there has been a history of infertility
* Patients who are HCV and HBV negative

Exclusion Criteria

* patients who have a calculated GFR (Nankivell formula) of less than 30mL/min at baseline
* Patients who are recipients of multiple organ transplants
* Patients who are recipients of dual kidney transplants
* Patients with panel reactive antibodies >50% at transplant
* Patients with a known hypersensitivity to tacrolimus,EC-MPS or basiliximab at baseline
* Patients with a known malignancy or a history of malignancy, other than successfully treated non-metastatic basal or squamous cell carcinoma of the skin
* Patients who are HIV positive at study entry
* Patients who have received a kidney from a HCV positive or HBV positive donor
* Patients with signs of active immune process on graft biopsy at baseline
* Patients with polyoma (BK or JC)
* Patients with operative or technical failure

Exclusion Criteria:

-

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2007-04; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
To compare the annualised change in GFR (delta GFR) at three and twelve months after baseline.

SECONDARY OUTCOMES:
To demonstrate that the efficacy of basiliximab compared to the efficacy of tacrolimus kis comparable in the prevention of acute cellular rejection at 3 and 12 months after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: jean tchervenkov, MD, Principal Investigator — Royal Victoria Hospital, Canada
Locations (1):
- MUHC Royal Victoria Hospital, Montreal, Quebec, Canada